CLINICAL TRIAL: NCT00250367
Title: The Safety And Efficacy Of Risperdal� (Risperidone) Versus Placebo As Add-On Therapy To Mood Stabilizers In The Treatment Of The Manic Phase Of Bipolar Disorder
Brief Title: A Study of the Effectiveness and Safety of Risperidone Versus Placebo as add-on Therapy to Mood Stabilizers, in the Treatment of Manic Episodes Associated With Bipolar Disorder.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006058
Record Dates: First submitted 2005-11-04; First posted 2005-11-08 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2010-11

CONDITIONS: Bipolar Disorder; Manic Disorder
Keywords: risperidone; antipsychotic agents; bipolar disorders; manic episode
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of the study is to evaluate the effectiveness and safety of risperidone (an antipsychotic medication) versus placebo as add-on therapy to mood stabilizers, in the treatment of manic episodes associated with bipolar disorder.

DETAILED DESCRIPTION:
Risperidone, widely used in the treatment of schizophrenia, has been shown to be effective in the treatment of manic and mixed episodes associated with bipolar disorders. Antipsychotic drugs like risperidone have also been used as therapeutic agents in the treatment of patients who are not responsive to mood stabilizers alone. This is a randomized, double-blind study to evaluate the effectiveness and safety of risperidone compared with placebo, as an addition to mood stabilizing drugs, in the treatment of patients experiencing manic episodes associated with bipolar disorder. The study has two phases: a double-blind treatment phase (3 weeks) and an open-label phase (10 weeks). To participate in the study, patients must be in-patients for a minimum of the first 4 days of double-blind treatment. During the double-blind treatment phase, patients receive risperidone or placebo tablets to be taken once a day at gradually increasing doses at investigator's discretion, up to a maximum dose of 6 mg/day, while continuing their treatment with a mood stabilizer (lithium, valproate, or carbamazepine). In the open-label phase, therapy with a mood stabilizer continues, and all patients receive risperidone with dosage gradually adjusted to achieve optimal effectiveness. The primary measure of effectiveness is the change in Young Mania Rating Scale (YMRS) total score from baseline to end of double-blind treatment. Additional efficacy measures include the Brief Psychiatric Rating Scale (BPRS), the Clinical Global Impression (CGI), (which evaluates the change in severity of the disorder), and the Hamilton Depression Rating Scale (HAMD). Safety assessments include the incidence of adverse events throughout the study; measurement of vital signs (pulse and blood pressure) and evaluation of the presence and severity of extrapyramidal symptoms by the Extrapyramidal Symptom Rating Scale (ESRS) at specified intervals; and clinical laboratory tests (hematology, biochemistry, urinalysis) before study initiation, at completion of the double-blind treatment, and at the end of the study. The study hypothesis is that daily treatment with risperidone as add-on therapy provides better effectiveness than the addition of placebo, as measured by Young Mania Rating Scale scores, in the treatment of the manic phase of bipolar disorder. Risperidone 1 mg tablets, taken orally, once daily; Doses of 2 mg on Days 1 and 2, up to 4 mg on Days 3 and 4, and up to 6 mg (maximum dose) on Days 5 through 21. Same dose maintained through the 10 week open-label phase. Gradual dose adjustments are allowed to achieve optimal effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for mania with a score >=20 on the Young Mania Rating Scale (YMRS). (Patients with symptoms of depression are eligible)
* diagnosis of Bipolar Disorder according to Diagnostic and Statistical Manual of Mental Diseases, 4th edition (DSM-IV)
* receiving treatment with a mood stabilizer for a minimum of 2 weeks prior to study initiation, or beginning therapy with a mood stabilizer prior to treatment with study medication
* patients medically stable on the basis of physical examination, medical history and electrocardiogram results.

Exclusion Criteria:

* Other Axis I DSM-IV diagnosis (except nicotine or caffeine dependence)
* history of alcohol or drug abuse or dependence within 3 months of starting the study
* seizure disorder requiring medication
* known sensitivity to risperidone, lithium, valproate or carbamazepine
* pregnant or nursing females, or those lacking adequate contraception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 1997-10; Study Completion 1999-11 (Actual)

PRIMARY OUTCOMES:
Change in Young Mania Rating Scale (YMRS) total score from baseline to end of double-blind treatment

SECONDARY OUTCOMES:
Changes from baseline to end of double-blind treatment in Brief Psychiatric Rating Scale (BPRS), Clinical Global Impression (CGI) - severity, and Hamilton Depression Rating Scale (HAMD); incidence of adverse events throughout study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.

REFERENCES:
- [Result] Yatham LN, Grossman F, Augustyns I, Vieta E, Ravindran A. Mood stabilisers plus risperidone or placebo in the treatment of acute mania. International, double-blind, randomised controlled trial. Br J Psychiatry. 2003 Feb;182:141-7. doi: 10.1192/bjp.182.2.141. PMID 12562742